CLINICAL TRIAL: NCT02934256
Title: Icotinib Hydrochloride Tablets Study for Patients With Neurofibromatosis Type 2 (NF2) and NF2-Related Tumors
Brief Title: Icotinib Study for Patients With Neurofibromatosis Type 2 (NF2) and NF2-Related Tumors
Acronym: Icotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Li Peng (Other)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Li Peng, principal investigator, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tian-drug-neuro002
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Vestibular Schwannoma; Neurofibromatosis Type 2
Keywords: Neurofibromatosis Type 2; Vestibular Schwannoma; Other NF2-related tumors
MeSH Terms: conditions — Neuroma, Acoustic; Neurofibromatosis 2 | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib，treatment effect evaluation (Experimental): Patients use Icotinib hydrochloride tablets during the course of treatment. The drug dosage is 125mg/m3/d. Every course of treatment lasts three months. Patients are designed to receive total four courses of treatment if there is no disease progression.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Method of drug administration:oral; Dosage: 125mg/m3/d; Course of treatment: 3 months;Total four treatment courses.
  Other Names: Icotinib Hydrochloride Tablets

SUMMARY:
1)Preliminarily evaluate the treatment effect of Icotinib Hydrochloride Tablets on NF2; 2)Preliminarily evaluate the safety and the patient's tolerance of the treatment of Icotinib; 3)Provide an objective basis for an enlarged randomized double-blind trial.

DETAILED DESCRIPTION:
Neurofibromatosis type 2 (NF2) is a hereditary tumor predisposition syndrome caused by mutations in the NF2 tumor suppressor gene. Individuals with NF2 have a higher likelihood to develop multiple nervous system tumors, including schwannomas, meningiomas, and ependymomas. The hallmark of NF2 is bilateral vestibular schwannomas. Historically, most NF2 patients experience complete hearing loss either from tumor progression or after treatment of the tumors with surgery or radiation. Effective treatments are urgently needed for NF2 patients with progressive hearing loss because hearing loss is associated with impairment in social, emotional,and communication function and with increased depression.

Previous studies of NF2 patients treated with Erlotinib suggested that inhibition of epidermal growth factor receptor (EGFR) could result in hearing improvement and reduction in tumor size.

Much evidence implicates human epidermal growth factor (HER) receptors in vestibular schwannoma growth.Some studies have demonstrated that Merlin, the NF2 gene protein product, controls surface availability of the EGFR, ErbB2, and ErbB3 receptors in human and Drosophila models. Besides, cell culture models of mouse embryo fibroblasts (MEFs) support the role of EGFR in NF2-associated tumorigenesis. Nf2-deficient cells in culture lack contact-dependent inhibition of growth and continue to grow in confluent cultures. This effect appears to be mediated by EGFR signaling. Treatment of Nf2-deficient cells with EGFR inhibitors such as gefitinib can restore contact-dependent inhibition, suggesting that this class of drugs might be useful for NF2 patients with progressive vestibular schwannomas. In this way, Icotinib can inhibit the nutrition of the tumor and decrease the tumor's growth and metastasis. Based on these studies, we perform this clinical trial to known the treatment effect and tolerability of Icotinib on NF2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at the age of 16-50
2. Patients must meet the diagnostic criteria for NF2, with bilateral acoustic neuroma and other central nervous system tumors
3. Patients must not be treated with other drugs or radiation therapy recently
4. Patients should live in Beijing or nearby and can be treated in hospital
5. Patients must be healthy and not be seriously allergic with biological agents
6. Patients must join the clinical trial voluntarily, with good compliance, cooperate with the researchers well, sign a written informed consent.

Exclusion Criteria:

1. Treated with other drugs, surgery or radiation therapy recently
2. Brainstem is compressed seriously, with hydrocephalus, need to be treated with surgery in short time
3. Being pregnant or try to get pregnant, lactating women
4. With acute or chronic infectious diseases
5. With heart diseases, cardiac dysfunction or abnormal ECG
6. With uncontrolled neural or mental diseases, poor compliance
7. Not available for enhanced MRI
8. Take part in any other clinical trial
9. With other conditions that are considered not suitable for this clinical trial.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in volume of tumour after every course of the treatment | Baseline,Month 3,Month 6,Month 9,Month 12
  Patients in this clinical trial would receive MRI test to evaluate the volume of tumour after every course of the treatment.

SECONDARY OUTCOMES:
Change from Baseline in hearing ability after every course of the treatment | Baseline,Month 3,Month 6,Month 9,Month 12
  Patients' hearing ability would be tested after every course of the treatment.

OTHER OUTCOMES:
Change from baseline in QOL(quality of life) score after every course of the treatment | Baseline,Month 3,Month 6,Month 9,Month 12
  Patients' QOL(quality of life) would be evaluated after every course of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pinan Liu, Study Director — Beijing Tiantan Hospital; Fu Zhao, Principal Investigator — Beijing Neurosurgical Institute
Locations (2):
- China (2):
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Undecided